CLINICAL TRIAL: NCT06411041
Title: Effects of a Combined Program of Pelvic Floor Muscle Training and Yoga on Relieving Genitourinary Symptoms, and Improving Sexual Function and Quality of Life in Asian Women With Breast Cancer
Brief Title: Effects of a Combined Program of Pelvic Floor Muscle Training and Yoga
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yuan-Mei Liao, RN, PhD, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24MMHIS120e
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Genitourinary Symptoms; Sexual Function; Quality of Life
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Intervention Model Description: The experimental group will receive regular care and a 12-week program of pelvic floor muscle training (PFMT) and yoga. The control group will receive regular care.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will not be informed about the group of the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The experimental group will receive regular care and a 12-week program of pelvic floor muscle training (PFMT) and yoga
  Interventions: Behavioral: Pelvic Floor Muscle Training (PFMT) and yoga
- Control group (No Intervention): The control group will receive regular care

INTERVENTIONS:
Behavioral: Pelvic Floor Muscle Training (PFMT) and yoga — The experimental group participants will be instructed to perform the practice session four days a week. The four days per week practice times (PFMT 15 minutes/day; yoga 40 minutes/day.) will result in weekly practice times for pelvic floor muscle training (PFMT) of 60 minutes and for yoga of ≥150 minutes.
  Arms: Intervention group

SUMMARY:
This study aims to examine the effects of Pelvic Floor Muscle Training (PFMT) combined with yoga on relieving genitourinary symptoms, symptom-related quality of life, and improving sexual function in women with breast cancer. This study is a parallel randomized study with two groups. Women will be assigned to the experimental or control group by using the block randomization method. The experimental group will receive regular care and a 12-week program of PFMT and yoga. The control group will receive regular care. We collect relevant data from both groups at baseline and 4, 8, 12, and 24 weeks after baseline during the study period.

DETAILED DESCRIPTION:
This study will be conducted with the approval obtained from the Institutional Review Board (IRB) of MacKay Memorial Hospital. This parallel-two-group randomized experimental study including an experimental group and a control group examines the effects of pelvic floor muscle training (PFMT) combined with yoga on genitourinary symptoms, symptom-related quality of life, and sexual function. A sample of women with breast cancer experiencing ≥1 genitourinary symptom(s) will be recruited and assigned to an experimental group or a control group by using the block randomization method. The experimental group will receive regular care and a 12-week program of PFMT and yoga. We will provide the experimental group with 12 days of online group practice sections of PFMT and yoga (weekly 60-minute practice incudes yoga 40 minutes, PFMT 15 minutes, and reflection 5 minutes). We expect them to perform 36 days of home-based practice of PFMT and yoga with 3 days/week of yoga for 40 minutes and PFMT for 15 minutes. The control group will receive regular care and relevant educational materials after data collection. Information will be collected at five time points: baseline and 4, 8, 12, and 24 weeks after baseline. Generalized estimating equation procedures will be used to examine the effects of the intervention. We hypothesized that the experimental group will display more significant improvements in genitourinary symptoms, symptom-related influences, and sexual function than those shown in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-60 years
* Women with a confirmed diagnosis of breast cancer (Stages I-III) for ≥3 months
* Women who experience ≥1 genitourinary symptom(s)

Exclusion Criteria:

* Women with other types of cancer diagnoses (e.g., endometrial cancer and ovarian cancer)
* Women with inadequately managed chronic conditions (e.g., an individual with diabetes having HbA1c level >7%)

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women who aged 20-60 years, with a confirmed diagnosis of breast cancer (Stages I-III) for ≥3 months, and experience ≥1 genitourinary symptom(s)
Enrollment: 90 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Vulvovaginal Symptoms | Baseline
  The 21-item Chinese version of the Vulvovaginal Symptoms Questionnaire (C-VSQ) comprises four subscales to assess vulvovaginal symptoms experienced during the past week (Items 1-7), and symptom-related influences (Emotions Items 8-11; Life-impact Items 12-15, and Sexual-impact Items 16, 18-21). The response options for all items are "Yes" (1 point) and "No" (0 point). Subscale scores are the sum of the scores for the items included in that subscale. The C-VSQ total score is the sum of three subscale scores (0-15 points) or four subscale scores (0-20 points for sexually active women). A higher C-VSQ total score indicates experiencing greater severity of vulvovaginal symptoms and symptom-related influences.
Vulvovaginal Symptoms | 4 weeks after baseline
  The 21-item Chinese version of the Vulvovaginal Symptoms Questionnaire (C-VSQ) comprises four subscales to assess vulvovaginal symptoms experienced during the past week (Items 1-7), and symptom-related influences (Emotions Items 8-11; Life-impact Items 12-15, and Sexual-impact Items 16, 18-21). The response options for all items are "Yes" (1 point) and "No" (0 point). Subscale scores are the sum of the scores for the items included in that subscale. The C-VSQ total score is the sum of three subscale scores (0-15 points) or four subscale scores (0-20 points for sexually active women). A higher C-VSQ total score indicates experiencing greater severity of vulvovaginal symptoms and symptom-related influences.
Vulvovaginal Symptoms | 8 weeks after baseline
  The 21-item Chinese version of the Vulvovaginal Symptoms Questionnaire (C-VSQ) comprises four subscales to assess vulvovaginal symptoms experienced during the past week (Items 1-7), and symptom-related influences (Emotions Items 8-11; Life-impact Items 12-15, and Sexual-impact Items 16, 18-21). The response options for all items are "Yes" (1 point) and "No" (0 point). Subscale scores are the sum of the scores for the items included in that subscale. The C-VSQ total score is the sum of three subscale scores (0-15 points) or four subscale scores (0-20 points for sexually active women). A higher C-VSQ total score indicates experiencing greater severity of vulvovaginal symptoms and symptom-related influences.
Vulvovaginal Symptoms | 12 weeks after baseline
  The 21-item Chinese version of the Vulvovaginal Symptoms Questionnaire (C-VSQ) comprises four subscales to assess vulvovaginal symptoms experienced during the past week (Items 1-7), and symptom-related influences (Emotions Items 8-11; Life-impact Items 12-15, and Sexual-impact Items 16, 18-21). The response options for all items are "Yes" (1 point) and "No" (0 point). Subscale scores are the sum of the scores for the items included in that subscale. The C-VSQ total score is the sum of three subscale scores (0-15 points) or four subscale scores (0-20 points for sexually active women). A higher C-VSQ total score indicates experiencing greater severity of vulvovaginal symptoms and symptom-related influences.
Vulvovaginal Symptoms | 24 weeks after baseline
  The 21-item Chinese version of the Vulvovaginal Symptoms Questionnaire (C-VSQ) comprises four subscales to assess vulvovaginal symptoms experienced during the past week (Items 1-7), and symptom-related influences (Emotions Items 8-11; Life-impact Items 12-15, and Sexual-impact Items 16, 18-21). The response options for all items are "Yes" (1 point) and "No" (0 point). Subscale scores are the sum of the scores for the items included in that subscale. The C-VSQ total score is the sum of three subscale scores (0-15 points) or four subscale scores (0-20 points for sexually active women). A higher C-VSQ total score indicates experiencing greater severity of vulvovaginal symptoms and symptom-related influences.

SECONDARY OUTCOMES:
Urinary symptoms | Baseline
  We investigated eight common urinary symptoms using the lower urinary tract symptoms (LUTS) subscale. The LUTS subscale investigates (a) urinary incontinence, (b) increased daytime urinary frequency, (c) urgency, (d) nocturia, (e) intermittent stream/intermittency, (f) slow stream, (g) hesitancy, and (h) a feeling of incomplete emptying. A higher total LUTS score (Range 0-11) indicates that a woman experiences a greater number of different types of urinary symptoms.
Urinary symptoms | 4 weeks after baseline
  We investigated eight common urinary symptoms using the lower urinary tract symptoms (LUTS) subscale. The LUTS subscale investigates (a) urinary incontinence, (b) increased daytime urinary frequency, (c) urgency, (d) nocturia, (e) intermittent stream/intermittency, (f) slow stream, (g) hesitancy, and (h) a feeling of incomplete emptying. A higher total LUTS score (Range 0-11) indicates that a woman experiences a greater number of different types of urinary symptoms.
Urinary symptoms | 8 weeks after baseline
  We investigated eight common urinary symptoms using the lower urinary tract symptoms (LUTS) subscale. The LUTS subscale investigates (a) urinary incontinence, (b) increased daytime urinary frequency, (c) urgency, (d) nocturia, (e) intermittent stream/intermittency, (f) slow stream, (g) hesitancy, and (h) a feeling of incomplete emptying. A higher total LUTS score (Range 0-11) indicates that a woman experiences a greater number of different types of urinary symptoms.
Urinary symptoms | 12 weeks after baseline
  We investigated eight common urinary symptoms using the lower urinary tract symptoms (LUTS) subscale. The LUTS subscale investigates (a) urinary incontinence, (b) increased daytime urinary frequency, (c) urgency, (d) nocturia, (e) intermittent stream/intermittency, (f) slow stream, (g) hesitancy, and (h) a feeling of incomplete emptying. A higher total LUTS score (Range 0-11) indicates that a woman experiences a greater number of different types of urinary symptoms.
Urinary symptoms | 24 weeks after baseline
  We investigated eight common urinary symptoms using the lower urinary tract symptoms (LUTS) subscale. The LUTS subscale investigates (a) urinary incontinence, (b) increased daytime urinary frequency, (c) urgency, (d) nocturia, (e) intermittent stream/intermittency, (f) slow stream, (g) hesitancy, and (h) a feeling of incomplete emptying. A higher total LUTS score (Range 0-11) indicates that a woman experiences a greater number of different types of urinary symptoms.

OTHER OUTCOMES:
Sexual function | Baseline
  The 19-item Female Sexual Function Index (FSFI) consists of six domains: sexual desire (Items 1-2), subjective arousal (Items 3-6), lubrication (Items 7-10), orgasm (Items 11-13), satisfaction (Items 14-16), and pain (Items 17-19). The total score is the sum of all the item scores. A higher FSFI total score indicates better overall sexual functioning.
Sexual function | 4 weeks after baseline
  The 19-item Female Sexual Function Index (FSFI) consists of six domains: sexual desire (Items 1-2), subjective arousal (Items 3-6), lubrication (Items 7-10), orgasm (Items 11-13), satisfaction (Items 14-16), and pain (Items 17-19). The total score is the sum of all the item scores. A higher FSFI total score indicates better overall sexual functioning.
Sexual function | 8 weeks after baseline
  The 19-item Female Sexual Function Index (FSFI) consists of six domains: sexual desire (Items 1-2), subjective arousal (Items 3-6), lubrication (Items 7-10), orgasm (Items 11-13), satisfaction (Items 14-16), and pain (Items 17-19). The total score is the sum of all the item scores. A higher FSFI total score indicates better overall sexual functioning.
Sexual function | 12 weeks after baseline
  The 19-item Female Sexual Function Index (FSFI) consists of six domains: sexual desire (Items 1-2), subjective arousal (Items 3-6), lubrication (Items 7-10), orgasm (Items 11-13), satisfaction (Items 14-16), and pain (Items 17-19). The total score is the sum of all the item scores. A higher FSFI total score indicates better overall sexual functioning.
Sexual function | 24 weeks after baseline
  The 19-item Female Sexual Function Index (FSFI) consists of six domains: sexual desire (Items 1-2), subjective arousal (Items 3-6), lubrication (Items 7-10), orgasm (Items 11-13), satisfaction (Items 14-16), and pain (Items 17-19). The total score is the sum of all the item scores. A higher FSFI total score indicates better overall sexual functioning.
Quality of life and distress associated with pelvic floor symptoms | Baseline
  The 20-item Pelvic Floor Distress Inventory-20 (PFDI-20) consists of three sections: Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6; Items 1-6), Colorectal-Anal Distress Inventory (CRAD-8; Items 7-14), and Urinary Distress Inventory 6 (UDI-6; Items 15-20). The total score ranges from 0-300, and a higher PFDI-20 total score indicates more severe influences associated with pelvic floor symptoms.
Quality of life and distress associated with pelvic floor symptoms | 4 weeks after baseline
  The 20-item Pelvic Floor Distress Inventory-20 (PFDI-20) consists of three sections: Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6; Items 1-6), Colorectal-Anal Distress Inventory (CRAD-8; Items 7-14), and Urinary Distress Inventory 6 (UDI-6; Items 15-20). The total score ranges from 0-300, and a higher PFDI-20 total score indicates more severe influences associated with pelvic floor symptoms.
Quality of life and distress associated with pelvic floor symptoms | 8 weeks after baseline
  The 20-item Pelvic Floor Distress Inventory-20 (PFDI-20) consists of three sections: Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6; Items 1-6), Colorectal-Anal Distress Inventory (CRAD-8; Items 7-14), and Urinary Distress Inventory 6 (UDI-6; Items 15-20). The total score ranges from 0-300, and a higher PFDI-20 total score indicates more severe influences associated with pelvic floor symptoms.
Quality of life and distress associated with pelvic floor symptoms | 12 weeks after baseline
  The 20-item Pelvic Floor Distress Inventory-20 (PFDI-20) consists of three sections: Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6; Items 1-6), Colorectal-Anal Distress Inventory (CRAD-8; Items 7-14), and Urinary Distress Inventory 6 (UDI-6; Items 15-20). The total score ranges from 0-300, and a higher PFDI-20 total score indicates more severe influences associated with pelvic floor symptoms.
Quality of life and distress associated with pelvic floor symptoms | 24 weeks after baseline
  The 20-item Pelvic Floor Distress Inventory-20 (PFDI-20) consists of three sections: Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6; Items 1-6), Colorectal-Anal Distress Inventory (CRAD-8; Items 7-14), and Urinary Distress Inventory 6 (UDI-6; Items 15-20). The total score ranges from 0-300, and a higher PFDI-20 total score indicates more severe influences associated with pelvic floor symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Mei Liao, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Data are available on request due to privacy and ethical restrictions.
Supporting Information: SAP
Time Frame: Baseline and 4, 8, 12 weeks after baseline
Access Criteria: Data are available on request due to privacy and ethical restrictions.